CLINICAL TRIAL: NCT00457925
Title: An Open-label, Two Period Study to Determine the Excretion Balance and Pharmacokinetics of [14C]-GSK221149A, Administered as Single Doses of an Oral Solution and an Intravenous Infusion to Healthy Female Volunteers
Brief Title: Absorption, Distribution, Metabolism And Excretion Study For GSK221149A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTA105101
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Obstetric Labour, Premature; Premature Labor
Keywords: absorption,; metabolism,; excretion; distribution,
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — GSK221149A

INTERVENTIONS:
Drug: GSK221149A

SUMMARY:
This is a phase one study investigating the absorption, distribution, metabolism and excretion of GSK221149A in six healthy women of non-child bearing potential.

ELIGIBILITY:
Inclusion criteria:

* Healthy adult, non-smoking females
* Aged between 30 - 55 years old, and BMI of between 19 and 32
* Not of child-bearing potential

Exclusion criteria:

* No clinically significant findings on clinical examination, medical examination and blood tests.
* Radiation exposure over previous 3 years is greater than 10mSv
* History of bleeding or gastric problems

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6
Dates: Start 2006-10

PRIMARY OUTCOMES:
Urinary and fecal cumulative excretion as a percentage of the total radioactive dose administered over time. Collection of plasma, urine and fecal samples for assessment of metabolites. Samples are collected for approximately 7 days (or longer).

SECONDARY OUTCOMES:
Clinical Safety data. PK parameters of GSK221149A and drug-related material (radioactivity) in plasma following oral and intravenous dosing. Samples are collected for approximately seven days (or longer) following dosing.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States